CLINICAL TRIAL: NCT02194725
Title: Where Does Hope Fit In? The Relationship Between Hope, Uncertainty, and Coping Efficacy in Mothers of Children With Duchenne/Becker Muscular Dystrophy
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999914149; 14-HG-N149
Record Dates: First submitted 2014-07-16; First posted 2014-07-18 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2017-07-07

CONDITIONS: Stress
Keywords: Stress and Coping Model; Coping

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional

SUMMARY:
Background:

- Children with Duchenne/Becker Muscular Dystrophy (DBMD) slowly lose muscle function. They usually die at a young age. Some mothers adapt to the demands of caring for a child with this disease better than others. Studies show that a person s hope may positively affect how they cope and adapt. Researchers want to find out more about this. They want to develop ways to improve caregivers overall wellness.

Objective:

- To study the relationships between uncertainty, hope, and coping ability in mothers of children with DBMD.

Eligibility:

- Women in the United States 18 years and older. They must be biological mothers of a living child with DBMD and be able to answer a survey in English.

Design:

* This study is part of a larger study that examines the well-being of mothers with sons who have DBMD.
* Participants will take a questionnaire. The questionnaire can be done on paper or on a computer. It will take 30 45 minutes to complete.
* The questionnaire will include basic demographic questions about the participant and the child. There will also be questions about how the participant copes with the stress and uncertainty of DBMD.
* For most of the questions, participants will rate their feelings on a scale. There will also be four open-ended questions.

DETAILED DESCRIPTION:
The proposed study aims to examine the relationships between maternal uncertainty, hope, and coping efficacy in mothers of children with Duchenne/Becker Muscular Dystrophy (DBMD). DBMD is described as a complex chronic condition causing challenges exemplified by both chronic and terminal illnesses. Parental adaptation to a child s DBMD diagnosis is multifaceted due to the evolution of the disease and uncertain timing of the progressive losses the child and family face. In addition to prognostic uncertainty associated with DBMD, there is uncertainty about the management of the condition, future and reproductive planning, the family s social connections, and the existential meaning of the child s life. It is not fully understood how mothers of children with DBMD appraise, cope with, and ultimately adapt to their child s condition in light of this uncertainty. While high degrees of perceived uncertainty may be seen as a threat to coping and adaptation, there is evidence that caregivers may find benefits in uncertainty. The theoretical literature suggests that a person s hope may influence the appraisal of uncertainty, as well as have therapeutic value in positively affecting coping and ultimately, adaptation. This study s conceptual framework is based on an integrated model from Lazarus and Folkman s Transactional Model of Stress and Coping, Mishel s Perceived Uncertainty in Illness Theory, and Dufault and Martocchio s Model of Hope. The proposed study uses a cross-sectional research design to explore the relationships between maternal uncertainty, hope, and coping efficacy and is nested within a larger longitudinal study designed to examine the predictors of wellbeing among mothers of boys with DBMD. In addition, open-ended questions will be used to describe the uncertainty the mothers perceive and the impact uncertainty has had on their life. Participants were recruited through the DuchenneConnect registry, Parent Project Muscular Dystrophy (PPMD), and Cincinnati Children s Hospital Medical Center Neuromuscular Clinic. Additional mothers will be recruited through the DuchenneConntect registry, PPMD, and the Muscular Dystrophy Association.

ELIGIBILITY:
* INCLUSION CRITERIA:

Participants will be biological mothers of a living child with Duchenne or Becker muscular dystrophy living in the United States, who are 18 years or older and able to answer a survey in English.

Participants will be asked to disclose their child's diagnosis but no screening evaluation will be required.

EXCLUSION CRITERIA:

Participants unable to answer a survey in English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 228 (Actual)
Dates: Start 2014-07-06; Primary Completion 2015-04-20 (Actual); Study Completion 2017-07-07 (Actual)

PRIMARY OUTCOMES:
Coping Efficacy | Current

SECONDARY OUTCOMES:
Uncertainty | Current
Adaptation | Current

CONTACTS AND LOCATIONS:
Overall Officials: Barbara B Biesecker, Principal Investigator — National Human Genome Research Institute (NHGRI)
Locations (1):
- National Human Genome Research Institute (NHGRI), 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ballew SH, Hannum SM, Gaines JM, Marx KA, Parrish JM. The role of spiritual experiences and activities in the relationship between chronic illness and psychological well-being. J Relig Health. 2012 Dec;51(4):1386-96. doi: 10.1007/s10943-011-9498-0. PMID 21604081
- [Background] Bedard M, Molloy DW, Squire L, Dubois S, Lever JA, O'Donnell M. The Zarit Burden Interview: a new short version and screening version. Gerontologist. 2001 Oct;41(5):652-7. doi: 10.1093/geront/41.5.652. PMID 11574710
- [Background] Biesecker BB, Erby LH, Woolford S, Adcock JY, Cohen JS, Lamb A, Lewis KV, Truitt M, Turriff A, Reeve BB. Development and validation of the Psychological Adaptation Scale (PAS): use in six studies of adaptation to a health condition or risk. Patient Educ Couns. 2013 Nov;93(2):248-54. doi: 10.1016/j.pec.2013.05.006. Epub 2013 Aug 28. PMID 23993396